CLINICAL TRIAL: NCT06835621
Title: Comparison of Functional Recovery Between Restricted Inverse Kinematic Alignment and Adjusted Mechanical Alignment With Robotic-assisted Unilateral Total Knee Arthroplasty. A Randomized Controlled Trial.
Brief Title: Comparison of Functional Recovery Between Restricted Inverse Kinematic Alignment and Adjusted Mechanical Alignment With Robotic-assisted Unilateral Total Knee Arthroplasty.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Krit Boontanapibul, Associate Professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTU-EC-OT-0-240/67
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: OA Knee; TKA
Keywords: Osteoarthritis (OA) of the Knee; OA knee; MAKO; Kinematic alignment; Mechanical alignment; Restricted Kinematic alignment; Inversed Kinematic alignment; Inversed Restricted Kinematic alignment; Robotic assist Total Knee Arthroplasty; Adjusted mechanical alignment
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Restricted inverse kinematic alignment
  Interventions: Procedure: Restricted inverse kinematic alignment Total Knee Arthroplasty
- Group 2 (Active Comparator): Adjusted mechanical alignment
  Interventions: Procedure: Adjusted Mechanical alignment Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Restricted inverse kinematic alignment Total Knee Arthroplasty — Restricted inverse kinematic alignment (restricted iKA) total knee arthroplasty is an alignment technique of total knee replacement surgery, aim to maintain the native coronal alignment within a HKA angle safe zone of 177° to 183°. This technique aims to 'resurface' the femur maintaining the native femoral joint line obliquity, with the flexion and extension gaps balanced by adjusting the tibial resection first. It is considered a more personalized approach because it aims to replicate the knee's pre-arthritic alignment and movement, believing that each patient's knee has a unique alignment.
  Other Names: Restricted kinematic alignment; rKA; Inverse kinematic alignment; iKA; Restricted iKA
  Arms: Group 1
Procedure: Adjusted Mechanical alignment Total Knee Arthroplasty — The adjusted Mechanical Alignment (aMA) technique is an adaptation of the conventional MA technique but with undercorrection of constitutional coronal deformity, within a limit of ± 3°. The femoral resection is adjusted to preserve mild constitutional deformity and/or reduce more severe deformity while leaving the tibial component mechanically aligned. The tibial component was positioned with the aim to be perpendicular (90°) to the mechanical tibial axis.
  Other Names: aMA
  Arms: Group 2

SUMMARY:
The goal of this clinical trial is to learn if restricted inverse kinematic alignment total knee arthroplasty (restricted iKA TKA) improves functional recovery compared to adjusted mechanical alignment total knee arthroplasty (aMA TKA) in patients undergoing unilateral robotic-assisted total knee arthroplasty by comparing performance-based outcome, 2-minute walk test (2MWT) as a primary outcome. This trial will also assess other outcomes including satisfaction, patient-reported functional outcomes, range of motion, visual analog scale for pain and complication of both techniques. The main question aims to answer is:

In unilateral robotic-assisted total knee arthroplasty, dose Restricted iKA technique provide better postoperative performance-based outcome compared to aMA technique?

Researchers will compare restricted iKA and aMA technique to determine which technique offers better acceleration in functional recovery and patient satisfaction.

Participants will:

After randomization, participants will allocate to either restricted iKA or aMA technique for unilateral robotic-assisted total knee arthroplasty.

Attend follow-up visits for assessments of 2-minute walk test (Primary outcome), Time up and go test (TUG), VAS for pain, ROM and complete patient-reported functional outcome questionnaires regarding knee function and satisfaction at regular intervals.

DETAILED DESCRIPTION:
Nowadays, total knee arthroplasty (TKA) for the treatment of osteoarthritis patients generally aims to achieve a neutral alignment of the leg. This involves cutting the bones perpendicular to the mechanical axis in both the femur and tibia. This method is called mechanical alignment TKA (MA TKA), which is widely popular and is often considered the standard technique for TKA. It has shown satisfactory long-term outcomes. However, despite advancements in materials and surgical techniques, MA TKA still requires bone and soft tissue adjustments to correct alignment, which may involve releasing soft tissues. This can result in post-surgical pain or dissatisfaction, with up to 20% of patients reporting dissatisfaction despite improved knee pain compared to pre-surgery. Furthermore, 1 in 4 of these dissatisfied patients do not wish to undergo a revision surgery, as the MA TKA method is a "one-size-fits-all" approach that aims to achieve equal and parallel gaps between the femur and tibia components without respecting individual soft tissue balance and the original alignment of each patient's leg. However, adjusted mechanical alignment technique, an adaptation of conventional MA technique with under-correction of constitutional coronal deformity, within a limit of ± 3° (HKA -3° to 3) has been introduced according to the constitutional deformity and coronal plan alignment of the knee concept.

In 2006, Howell introduced kinematic alignment TKA (KA TKA) as an alternative, with the goal of restoring the patient's natural kinematic axis and reducing the incidence of pain related to TKA rather than focusing on equal medial and lateral joint line gap and neutral mechanical axis like in mechanical alignment technique. KA TKA is considered a more personalized approach because it aims to replicate the knee's pre-arthritic alignment and movement, believing that each patient's knee has a unique alignment. This approach has gained increasing interest in recent years, with studies reporting good short- to mid-term clinical outcomes. However, the KA technique is more complex because we cannot always know the pre-arthritic alignment of individual patients and measuring soft tissue tension remains imprecise.

Later, Dr. Pascal-André Vendittoli proposed the restricted kinematic alignment TKA (rKA TKA) technique to restore natural knee movement while avoiding excessive correction of coronal alignment by maintain the HKA axis within ± 3 degrees (safe zone). By maintaining some of the constitutional deformity, this technique reduces the need for excessive soft tissue or ligament releases. In 2020 Winnock et al, introduced the Inversed kinematic technique (iKA) or tibia-referenced technique by resurfacing the tibia with equal medial and lateral resections maintaining the native tibial joint line obliquity before distal femoral bone. When combines these KA principles with robotic-assisted TKA, enhancing the accuracy of soft tissue balancing and the overall effectiveness of the procedure.

In 2020, McEwen et al. compared the use of robotic-assisted KA with MA in the same patients who underwent bilateral knee surgery using different techniques. They found that clinical outcomes, including range of motion and knee scores, were not significantly different at any time point. However, Elbuluk conducted a similar comparison, specifically robotic-assisted (MAKO) KA versus MA, and found that the KA group had less pain and better knee scores, including a higher Forgotten Joint Score. Later, Abhari conducted a study comparing robotic-assisted (MAKO) restricted KA with non-robotic MA TKA and found that the robotic-assisted (MAKO) restricted KA group had superior clinical outcomes and knee scores, including the Forgotten Joint Score, KOOS, WOMAC, Knee Society Score, as well as greater patient satisfaction. However, there are still limited prospective RCTs that study differences in outcomes, especially performance-based outcomes between restricted inverse kinematic alignment (restricted iKA) versus adjusted mechanical alignment (aMA). Therefore, the researchers aim to conduct a study comparing the efficiency of performance-based outcomes as a primary focus, including patient-reported outcome questionnaires, ROM, VAS for postoperative pain, postoperative morphine consumption within 24 hours, postoperative lower limb alignment (HKA axis), operative time, blood loss, and complications. The goal is to further advance the development of knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 - 80 years old
* Diagnosed with primary OA knee and indicated for unilateral total knee arthroplasty with MAKO robotic-assisted knee replacement system
* ASA classification I-II

Exclusion Criteria:

* Valgus deformity
* KL grading > 3 on contralateral knee
* Unable or difficulty for walking due to comorbidities
* BMI > 40 kg/m2
* Previous knee surgery
* Infection around the knee

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
2-minute walk test | From enrollment (preoperative measurement) to the end of postoperative follow-up (2 years)
  The 2-minute walk test (2mwt) is a performance-based test that evaluates functional recovery after total knee arthroplasty (TKA) by measures the distance a person can walk in two minutes (meters) and has been validated as performance-based test with responsiveness properties. Being simple and easy to perform, it can be used routinely in clinical practice to evaluate functional recovery after TKA.

SECONDARY OUTCOMES:
Time up and go test | From enrollment (preoperative measurement) to the end of postoperative follow-up (2 years)
  The Timed Up and Go test (TUG) are simple, quick, and can be applied in a short time as part of the routine medical examination. They were shown to be reliable and valid tests in many patient groups including postoperative performance-based outcome for patients undergone TKA.
modified WOMAC scale for knee pain (Thai version) | From enrollment (preoperative measurement) to the end of postoperative follow-up (2 years)
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used questionnaire for assessing pain, stiffness, and functional limitation in patients with osteoarthritis, particularly in the knee and hip joints. The modified WOMAC scale adapts the original WOMAC to better suit specific populations or clinical settings. In this study, we use the modified WOMAC scale for knee pain Thai version to assess the pre and post operative functional outcome.
Thai version of the Forgotten Joint Score | From enrollment (preoperative measurement) to the end of postoperative follow-up (2 years)
  This score aims for evaluation of joint awareness in everyday life, which is one of the aspects to evaluate the outcome and the ability to forget the artificial joint, is claimed as the ultimate goal resulting in maximum patient satisfaction. The Thai language version of the FJS had high level of internal consistency and was proved to be a reliable tool for evaluating knee arthroplasty patients in Thailand. The low ceiling effect characteristic of the score can help the surgeon to detect small difference in the good and excellent outcomes after knee arthroplasty.
Oxford knee score | From enrollment (preoperative measurement) to the end of postoperative follow-up (2 years)
  The Oxford Knee Score (OKS) is a widely used patient-reported outcome measure designed to assess the function and quality of life of individuals with knee problems, particularly those undergoing knee surgery, such as total knee arthroplasty. It focuses specifically on how knee-related issues affect daily activities and overall well-being. (Thai version is available on the official website of the Oxford knee score website)
Range of Motion | From enrollment (preoperative measurement) to the end of postoperative follow-up (2 years)
  Preoperative and Postoperative active range of motion (ROM) will be recorded for evaluation of the knee ROM for both groups including flexion contracture (FC) or extension gap which may be presented as complication.
Hip knee ankle angle | From enrollment (preoperative measurement) and at 1-year postoperative follow-up.
  The hip knee ankle angle is radiographic measurement for determine the coronal alignment of the lower limbs. On a weight-bearing, full-length AP lower limb radiograph measuring 2 lines from center of the femoral head to the femoral intercondylar notch, while the latter from the tibial interspinous point to the tibial mid-plafond. The HKA is defined as the angle between these two lines.
Visual analog scale for Pain | From enrollment (preoperative measurement) to the end of postoperative follow-up (2 years)
  Each patient will be asked for Visual analog scale (VAS) for pain for the knee, which is the subjective patient reported pain rating from 0-10 either from numerical order or facial expression picture indicating 0 is the minimum or no pain and 10 is the maximum or the worst pain.
Morphine consumption | Postoperative interval of 24-72 hours
  Postoperative morphine consumption (mg) in the first 72 hours during hospital admission could reflect the need of strong opioid as the rescue analgesia after operation.
Complication | After surgery and up to 2 years
  Total knee arthroplasty-related complication e.g. surgical site infection, bleeding, wound complication, deep vein thrombosis, acute pulmonary embolism and implant failure.
Medial proximal tibial angle (MPTA) | From enrollment (preoperative measurement) and at 1-year postoperative follow-up.
  In whole leg AP weight baring film, measure the proximal medial angle formed between the tibial mechanical axis and the knee joint line of the tibia in the frontal plane.
Lateral distal femoral angle (LDFA) | From enrollment (preoperative measurement) and at 1-year postoperative follow-up.
  In whole leg AP weight baring film, it's defined as the lateral angle formed between the mechanical axis line of the femur and the knee joint line of the femur.
Joint line obliquity (JLO) | From enrollment (preoperative measurement) and at 1-year postoperative follow-up.
  Joint line obliquity (degrees) = MPTA + LDFA

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Thammasat University, Klongluang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elbuluk AM, Jerabek SA, Suhardi VJ, Sculco PK, Ast MP, Vigdorchik JM. Head-to-Head Comparison of Kinematic Alignment Versus Mechanical Alignment for Total Knee Arthroplasty. J Arthroplasty. 2022 Aug;37(8S):S849-S851. doi: 10.1016/j.arth.2022.01.052. Epub 2022 Jan 31. PMID 35093548
- [Background] McEwen PJ, Dlaska CE, Jovanovic IA, Doma K, Brandon BJ. Computer-Assisted Kinematic and Mechanical Axis Total Knee Arthroplasty: A Prospective Randomized Controlled Trial of Bilateral Simultaneous Surgery. J Arthroplasty. 2020 Feb;35(2):443-450. doi: 10.1016/j.arth.2019.08.064. Epub 2019 Sep 5. PMID 31591010
- [Background] Van Essen J, Stevens J, Dowsey MM, Choong PF, Babazadeh S. Kinematic alignment results in clinically similar outcomes to mechanical alignment: Systematic review and meta-analysis. Knee. 2023 Jan;40:24-41. doi: 10.1016/j.knee.2022.11.001. Epub 2022 Nov 17. PMID 36403396
- [Background] Blakeney WG, Vendittoli PA. Restricted Kinematic Alignment: The Ideal Compromise? 2020 Jul 1. In: Riviere C, Vendittoli PA, editors. Personalized Hip and Knee Joint Replacement [Internet]. Cham (CH): Springer; 2020. Chapter 17. Available from http://www.ncbi.nlm.nih.gov/books/NBK565760/ PMID 33347126
- [Background] Howell SM, Shelton TJ, Hull ML. Implant Survival and Function Ten Years After Kinematically Aligned Total Knee Arthroplasty. J Arthroplasty. 2018 Dec;33(12):3678-3684. doi: 10.1016/j.arth.2018.07.020. Epub 2018 Jul 31. PMID 30122435
- [Background] Vanlommel L, Vanlommel J, Claes S, Bellemans J. Slight undercorrection following total knee arthroplasty results in superior clinical outcomes in varus knees. Knee Surg Sports Traumatol Arthrosc. 2013 Oct;21(10):2325-30. doi: 10.1007/s00167-013-2481-4. Epub 2013 Apr 4. PMID 23552665
- [Background] Winnock de Grave P, Luyckx T, Claeys K, Tampere T, Kellens J, Muller J, Gunst P. Higher satisfaction after total knee arthroplasty using restricted inverse kinematic alignment compared to adjusted mechanical alignment. Knee Surg Sports Traumatol Arthrosc. 2022 Feb;30(2):488-499. doi: 10.1007/s00167-020-06165-4. Epub 2020 Jul 31. PMID 32737528
- [Background] Yang Y, Wang Y, Chen Y, Wang J, Lu B, Zhu W, Zhu J, Zhu C, Zhang X. Tracing the evolution of robotic-assisted total knee arthroplasty: a bibliometric analysis of the top 100 highly cited articles. J Robot Surg. 2023 Dec;17(6):2973-2985. doi: 10.1007/s11701-023-01742-4. Epub 2023 Oct 26. PMID 37882976
- [Background] Vendittoli PA, Martinov S, Blakeney WG. Restricted Kinematic Alignment, the Fundamentals, and Clinical Applications. Front Surg. 2021 Jul 20;8:697020. doi: 10.3389/fsurg.2021.697020. eCollection 2021. PMID 34355018
- [Background] Hirschmann MT, Becker R, Tandogan R, Vendittoli PA, Howell S. Alignment in TKA: what has been clear is not anymore! Knee Surg Sports Traumatol Arthrosc. 2019 Jul;27(7):2037-2039. doi: 10.1007/s00167-019-05558-4. Epub 2019 Jun 12. No abstract available. PMID 31190246
- [Background] Dossett HG, Estrada NA, Swartz GJ, LeFevre GW, Kwasman BG. A randomised controlled trial of kinematically and mechanically aligned total knee replacements: two-year clinical results. Bone Joint J. 2014 Jul;96-B(7):907-13. doi: 10.1302/0301-620X.96B7.32812. PMID 24986944
- [Background] Roth JD, Howell SM, Hull ML. Native Knee Laxities at 0 degrees , 45 degrees , and 90 degrees of Flexion and Their Relationship to the Goal of the Gap-Balancing Alignment Method of Total Knee Arthroplasty. J Bone Joint Surg Am. 2015 Oct 21;97(20):1678-84. doi: 10.2106/JBJS.N.01256. PMID 26491132
- [Background] Brar AS, Howell SM, Hull ML, Mahfouz MR. Does Kinematic Alignment and Flexion of a Femoral Component Designed for Mechanical Alignment Reduce the Proximal and Lateral Reach of the Trochlea? J Arthroplasty. 2016 Aug;31(8):1808-13. doi: 10.1016/j.arth.2016.01.040. Epub 2016 Feb 4. PMID 26923495
- [Background] Hiranaka T, Suda Y, Saitoh A, Tanaka A, Arimoto A, Koide M, Fujishiro T, Okamoto K. Current concept of kinematic alignment total knee arthroplasty and its derivatives. Bone Jt Open. 2022 May;3(5):390-397. doi: 10.1302/2633-1462.35.BJO-2022-0021.R2. PMID 35532356
- [Background] Nisar S, Palan J, Riviere C, Emerton M, Pandit H. Kinematic alignment in total knee arthroplasty. EFORT Open Rev. 2020 Aug 1;5(7):380-390. doi: 10.1302/2058-5241.5.200010. eCollection 2020 Jul. PMID 32818065